CLINICAL TRIAL: NCT07084753
Title: Comparison of Opioid-based Anesthesia, Opioid-free Anesthesia Based on Intravenous Drugs and Opioid-free Anesthesia With Thoracic Paravertebral Block, in Patients Undergoing Laparoscopic Gastric Bypass Surgery for Obesity
Brief Title: Non-opioid Anesthesia Based on Thoracic Paravertebral Block During Laparoscopic Sleeve Gastrectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IVO JURISIC (Other)
Responsible Party: Sponsor-Investigator, IVO JURISIC, MD, University Hospital Dubrava
Organization: University Hospital Dubrava (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023- 2301-08
Record Dates: First submitted 2025-06-23; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Obese Patients; Bariatric Surgical Pain; Bariatric Surgery (Sleeve Gastrectomy ); Non-Opioid Pain Management; PONV; Postoperative Analgesia; Postoperative Pain; Thoracic Paravertebral Block; Opioid Free Anesthesia
Keywords: thoracic paravertebral block; obese patients; bariatric surgery; sleeve gastrectomy; postoperative pain management; anesthesia recovery period; non-opioid anesthesia; recovery after bariatric surgery; TPVB; OFA based on thoracic paravertebral block; Visceral pain, Postoperative; Opioid based anesthesia; Opioid free anesthesia; OBA; OFA; Recovery Period, Anesthesia; Non-Opioid Pain Management; PONV; Postoperative analgesia; Postoperative pain; Bariatric Surgery, Pain; Opioid free anesthesia, dexmedetomidine, ketamine, lidocaine
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative; Visceral Pain; Pain | interventions — Levobupivacaine; Epinephrine; Dexmedetomidine; Ketamine; Sufentanil; Lidocaine; Metoclopramide; Thiethylperazine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Tthree groups of patients, each with 12 patients:
  1. opioid based aneshesia (OBA)
  2. opioid-free anesthesia with thoracic paravertebral block (TPVB)
  3. opioid free anesthesia with intravenous agents (OFA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Opioid based anesthesia (OBA) (Active Comparator): Premedication: pantoprazole 40 mg i.v. 1h before surgery. Following three-minute preoxygenation, sufentanil (5 to 15 micrograms), propofol (1 to 2 mg/kg ideal body weight), and rocuronium (0.8 to 1 mg/kg ideal body weight) are administered intravenously during induction of anesthesia. Anesthesia is sustained with sevoflurane maintained at 0.6-1.3 MAC. Sufentanil is added at the assessment of the anesthesiologist in the operating room. To prevent postoperative nausea and vomiting (PONV), patients receive intraoperatively dexamethasone (8 mg), ondansetron (4 mg), and metoclopramide (10 mg) intravenously. Intraoperative pain management includes metamizole (2.5 g) and acetaminophen (1 g). For pain levels of 4 or higher on a numerical rating scale (NRS), treatment options include metamizole (2.5 g), pethidine (25 to 100 mg), or tramadol (100 mg). For nausea and vomiting, intravenous doses of ondansetron or metoclopramide are provided as needed.
  Interventions: Drug: Sufentanil; Procedure: Opioid based Anesthesia; Drug: Metoclopramide 10mg; Drug: Ondasetron 4mg; Drug: Dexamethasone, 8 mg intravenously
- Opioid free anesthesia (OFA) based on lidocain, dexmedetomidine and S-ketamine (Active Comparator): Premedication: pregabalin 75 mg peroraly et pantoprazole 40mg i.v. A pre-prepared 50 ml syringe is utilized, containing 400 mcg of dexmedetomidine (4 ml), 50 mg of S-ketamine (2 ml), 400 mg of 2% lidocaine (20 ml), and 0.9% NaCl to a total volume of 40 ml. Anesthesia is commenced with the infusion from syringe 1 over a 10-minute period at a rate of 15 ml/hour. After this initial period, anesthetic induction is conducted using propofol at a dose of 1-2 mg/kg IBW and rocuronium at 0.8-1 mg/kg IBW. Anesthesia is sustained with sevoflurane maintained at 0.5-1 MAC, adjusted per BIS readings. The anesthetic mixture was maintained at a rate of 5-10 ml per hour adjusted according to the patient's blood pressure and pulse. Intraoperative pain management includes metamizole (2.5 g) and acetaminophen (1 g). To prevent nausea and vomiting, patients receive intraoperative dexamethasone 8 mg and thiethylperazine 6.5 mg intravenously.
  Interventions: Drug: Dexmedetomidin; Drug: ketamine; Drug: Lidocain; Procedure: Opioid free anesthesia, Opioid free anesthesia based on intravenous dexmedetomidine, ketamine and lidocainedexmedetomidine, ketamine and lidocaine; Drug: Thiethylperazine; Drug: Dexamethasone, 8 mg intravenously
- Opioid free anesthesia based on thoracic paravertebral block (TPVB) (Experimental): Premedication: pantoprazol 40mg i.v. Preoperative TPVB is executed at the Th5, Th7, and Th9 levels bilaterally. The skin at each level are infiltrated with 1.5 ml of 1% lidocaine. Subsequently, 10 ml of 0.33% levobupivacaine, combined with 1.33 mg of dexamethasone and 40 mcg of adrenaline, is injected at each level and flushed with 1 ml of 5% glucose. In the operating room a induction is carried out with propofol administered at a dosage of 2-2.5 mg/kg of ideal body weight (IBW) and rocuronium at 0.8-1 mg/kg of IBW. Anesthesia is maintained with an infusion of propofol at 100 mcg/kg of total body weight (TBW) per minute, with adjustments made to achieve a targeted BIS value between 40-60. Intraoperative pain management includes metamizole (2.5 g) and acetaminophen (1 g). Prophylaxis of PONV is dexamethasone 8 mg previously administered within the thoracic paravertebral block, with intraoperative administration of 10 mg metoclopramide.
  Completely opioid-free interventions.
  Interventions: Drug: Levobupivacaine; Drug: Dexamethasone contained in the solution for thoracic paravertebral block; Drug: Adrenaline; Procedure: Opioid free anesthesia based on thoracic paravertebral block; Device: Ultrasound guided thoracic paravertebral block; Device: Nerve stimulator for peripheral nerve blocks; Drug: Metoclopramide 10mg

INTERVENTIONS:
Drug: Levobupivacaine — Used in thoracic paravertebral block: 10 ml of 0.33% levobupivacaine, combined with 1.33 mg of dexamethasone and 40 mcg of adrenaline, is injected at each level (six levels, at the Th5, Th7, and Th9 levels bilaterally; a total of 200 mg of levobupivacaine, 8 mg of dexamethasone and 240 mcg of adrenaline).
  Arms: Opioid free anesthesia based on thoracic paravertebral block (TPVB)
Drug: Dexamethasone contained in the solution for thoracic paravertebral block — Used in thoracic paravertebral block: 10 ml of 0.33% levobupivacaine, combined with 1.33 mg of dexamethasone and 40 mcg of adrenaline, is injected at each level (six levels, at the Th5, Th7, and Th9 levels bilaterally; a total of 200 mg of levobupivacaine, 8 mg of dexamethasone and 240 mcg of adrenaline).
  Arms: Opioid free anesthesia based on thoracic paravertebral block (TPVB)
Drug: Adrenaline — Used in thoracic paravertebral block: 10 ml of 0.33% levobupivacaine, combined with 1.33 mg of dexamethasone and 40 mcg of adrenaline, is injected at each level (six levels, at the Th5, Th7, and Th9 levels bilaterally; a total of 200 mg of levobupivacaine, 8 mg of dexamethasone and 240 mcg of adrenaline).
  Arms: Opioid free anesthesia based on thoracic paravertebral block (TPVB)
Drug: Dexmedetomidin — A pre-prepared 50 ml syringe is utilized, containing 400 mcg of dexmedetomidine (4 ml), 50 mg of S-ketamine (2 ml), 400 mg of 2% lidocaine (20 ml), and 0.9% NaCl to a total volume of 40 ml. Anesthesia is commenced with the infusion from syringe 1 over a 10-minute period at a rate of 15 ml/hour. The anesthetic mixture was maintained at a rate of 5-10 ml per hour.
  Arms: Opioid free anesthesia (OFA) based on lidocain, dexmedetomidine and S-ketamine
Drug: ketamine — A pre-prepared 50 ml syringe is utilized, containing 400 mcg of dexmedetomidine (4 ml), 50 mg of S-ketamine (2 ml), 400 mg of 2% lidocaine (20 ml), and 0.9% NaCl to a total volume of 40 ml. Anesthesia is commenced with the infusion from syringe 1 over a 10-minute period at a rate of 15 ml/hour. The anesthetic mixture was maintained at a rate of 5-10 ml per hour.
  Arms: Opioid free anesthesia (OFA) based on lidocain, dexmedetomidine and S-ketamine
Drug: Lidocain — A pre-prepared 50 ml syringe is utilized, containing 400 mcg of dexmedetomidine (4 ml), 50 mg of S-ketamine (2 ml), 400 mg of 2% lidocaine (20 ml), and 0.9% NaCl to a total volume of 40 ml. Anesthesia is commenced with the infusion from syringe 1 over a 10-minute period at a rate of 15 ml/hour. The anesthetic mixture was maintained at a rate of 5-10 ml per hour.
  Arms: Opioid free anesthesia (OFA) based on lidocain, dexmedetomidine and S-ketamine
Drug: Sufentanil — Following three-minute preoxygenation, sufentanil (5 to 15 micrograms), propofol (1 to 2 mg/kg ideal body weight), and rocuronium (0.8 to 1 mg/kg ideal body weight) are administered intravenously during induction of anesthesia. Anesthesia is sustained with sevoflurane maintained at 0.6-1.3 MAC. Sufentanil is added at the assessment of the anesthesiologist in the operating room.
  Arms: Opioid based anesthesia (OBA)
Procedure: Opioid free anesthesia based on thoracic paravertebral block — Patients scheduled for laparoscopic sleeve gastrectomy will be anesthetized without the use of opioids, with general anesthesia and pain blockade using a thoracic paravertebral block
  Other Names: OFA based on TPVB
  Arms: Opioid free anesthesia based on thoracic paravertebral block (TPVB)
Procedure: Opioid based Anesthesia — Patients scheduled for laparoscopic sleeve gastrectomy will be anesthetized with opioids and general anesthesia
  Arms: Opioid based anesthesia (OBA)
Procedure: Opioid free anesthesia, Opioid free anesthesia based on intravenous dexmedetomidine, ketamine and lidocainedexmedetomidine, ketamine and lidocaine — Patients who are scheduled for laparoscopic gastrectomy will be anesthetized without the use of opioids and under general anesthesia, with analgesia by intravenous administration of dexmedetomidine, ketamine and lidocaine.
  Other Names: OFA
  Arms: Opioid free anesthesia (OFA) based on lidocain, dexmedetomidine and S-ketamine
Device: Ultrasound guided thoracic paravertebral block — Patients are positioned prone, with the identification of the 1st rib achieved using a convex XX Hz ultrasound probe. The left and right transverse processes of the 5th, 7th, and 9th thoracic vertebrae are marked accordingly. TPVB is executed in a paramedian sagittal oblique scan utilizing an in-plane needle insertion approach at the Th5, Th7, and Th9 levels bilaterally. An insulated echogenic needle, sized between 10-15 cm and 22-20 G, is employed. The skin and subcutaneous tissue at each level are infiltrated with 1.5 ml of 1% lidocaine.
  Ultrasound guidance combined with nerve stimulation (dual monitoring) is utilized at each corresponding paravertebral space. Verification of the paravertebral space is established through visualization of pleural displacement, as observed via the ultrasound probe following the injection of 1 ml of 5% glucose, as well as via a motor response at a current intensity of 0.3-0.5 mA.
  Other Names: Ultrasound guided TPVB
  Arms: Opioid free anesthesia based on thoracic paravertebral block (TPVB)
Device: Nerve stimulator for peripheral nerve blocks — During the application of the thoracic paravertebral block, verification of the distance of the insulated echogenic needle tip from the thoracic spinal nerve is monitored using via a motor response at a current intensity of 0.3-0.5 mA.
  Arms: Opioid free anesthesia based on thoracic paravertebral block (TPVB)
Drug: Metoclopramide 10mg — To prevent postoperative nausea and vomiting (PONV), patients receive dexamethasone (8 mg) and metoclopramide (10 mg) intraoperatively
  Arms: Opioid based anesthesia (OBA); Opioid free anesthesia based on thoracic paravertebral block (TPVB)
Drug: Ondasetron 4mg — To prevent postoperative nausea and vomiting (PONV), patients receive dexamethasone (8 mg), ondansetron (4 mg), and metoclopramide (10 mg) intraoperatively.
  Arms: Opioid based anesthesia (OBA)
Drug: Thiethylperazine — To prevent postoperative nausea and vomiting (PONV), patients receive dexamethasone (8 mg) and thiethylperazine (6.5 mg) intravenously.
  Arms: Opioid free anesthesia (OFA) based on lidocain, dexmedetomidine and S-ketamine
Drug: Dexamethasone, 8 mg intravenously — To prevent postoperative nausea and vomiting (PONV), patients receive intraoperatively dexamethasone (8 mg), ondansetron (4 mg), and metoclopramide (10 mg) intravenously.
  Arms: Opioid based anesthesia (OBA); Opioid free anesthesia (OFA) based on lidocain, dexmedetomidine and S-ketamine

SUMMARY:
Regional anesthesia is a technique in which a local anesthetic is injected near a nerve or spinal cord to block sensation, motor stimulation, and pain. In this study, an ultrasound-guided paravertebral block will be used, with careful consideration of all positive and negative factors and possible complications. A thoracic paravertebral block is performed by inserting a needle into the intercostal spaces on the back, approximately 4 cm lateral to the spine. Many studies support excellent pain control with this technique, during and after surgery in thoracic and abdominal surgery. Investigators aim to achieve faster patient mobility after surgery, rapid recovery of bowel function, reduced nausea and vomiting, and maximum pain control. The use of opioids, which can additionally cause respiratory suppression and drowsiness, is avoided.

At any time in case of need to switch from laparoscopic to open surgery, equally adequate anesthesia and postoperative analgesia are ensured without the need to change the approach to the same. In this study, the basic scientific assumption (hypothesis) of the researchers is that non-opioid anesthesia with thoracic paravertebral block provides adequate pain control during and long-term after the surgical procedure, without the side effects of opioid anesthesia.

The main goal of the study is to determine which type of anesthesia results in the best pain control and most significantly reduces complications of anesthesia and surgery in overweight patients who are scheduled for laparoscopic longitudinal gastrectomy and partial/total gastrectomy.

DETAILED DESCRIPTION:
Morbid obese patients scheduled for laparoscopic sleeve gastric resection need specific care during surgery and post-surgery. Postoperative pain management of these patients after this type of surgery is a challenge because of the high prevalence of nausea, vomiting, and higher risk of respiratory depression in obese patients, making the use of opioids undesirable. Various techniques have been used during and after surgery to control moderate to severe pain for early mobilization: OFA (opioid-free anesthesia) based on intravenous use of dexmedetomidine, ketamine, and lidocaine, or OBA (opioid-based anesthesia) in combination with regional anesthesia, to reduce the use of opioids. Regional anesthesia can be used as an additional modality of analgesia within OFA (opioid-free anesthesia) or opioid-based anesthesia (OBA), which either completely avoid the use of opioids or significantly reduce them. Investigators will compare opioid-based general anesthesia (OBA group) as the standard of anesthesia for bariatric surgery with intraoperative opioid- free anesthesia based on thoracic paravertebral block (TPVB group) and intraoperative opioid-free anesthesia based on intravenous dexmedetomidine, ketamine, and lidocaine (OFA group). The primary objective is to compare pain levels as measured by the 0-10 NRS and to compare opioid and analgesic consumption in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

-. patients with a prior history of treatment by a multidisciplinary obesity team scheduled for laparoscopic sleeve gastrectomy (LSG)

* body mass index of 30 kg/m² or greater
* patients classified as ASA status 2-3.

Exclusion Criteria:

* allergies to the intended medications
* patient refusal
* uncontrolled psychiatric disorders
* intracranial pathology
* cerebrovascular damage
* any factors impairing effective communication

Additional Exclusion Criteria:

1. For patients receiving thoracic paravertebral block (TPVB):

   - the presence of infection at the puncture site
2. For the OFA group:

   * 2nd or 3rd-degree atrioventricular block
   * bradycardia with a heart rate below 50 beats per minute
   * coronary artery disease,
   * cardiomyopathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
a) Postoperative pain levels measured by the 0-10 Numerical rating scale (NRS). b) Opioid analgesic consumption (Morphine milligram equivalents- MME). | 10 days
  1. Self-reported pain levels recorded at multiple time points:30 minutes post- surgery, every three hours for the first 24 hours, and three times daily for the following nine days. Zero indicates no pain, ten is the worst possible pain.
  2. Use of opioids (sufentanil, pethidine, tramadol) before, during and after surgery. Sufentanil in micrograms, pethidine and tramadol in milligrams. Values are converted into Morphine milligram equivalents (MME),

SECONDARY OUTCOMES:
a) Self-reported incidence of PONV after surgery. b) Time in the postoperative care unit (PACU) after surgery. c) Time to first mobilization after surgery. d) Time to fluid intake after surgery. | 10 days
  1. Recorded with a yes and no response.
  2. Measured in minutes (recorded in the patient's monitoring sheet).
  3. Measured in minutes (self-reported by the patient).
  4. Measured in minutes (self-reported by the patient).

CONTACTS AND LOCATIONS:
Overall Officials: IVO JURISIC, MD, Study Chair — University Hospital Dubrava
Locations (1):
- University Hospital Dubrava, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Yes
The plan is for the data to be made available after the study is completed and the article is published. Patients will be recorded by numbers and names will be omitted due to the General Data Protection Regulation (names will be known to the researcher). Access to the data will be possible upon request by a professional and with the approval of the University Hospital Dubrava Review Board.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The plan is for the data to be available after the study is completed and the article is published, within 365 days of the publication date.
Access Criteria: Access to the data will be possible upon request of experts to the researcher's e-mail and with the approval of the Review Board of the University Hospital Dubrava. When using data from this study for your own research or scientific work (presentation, article), it is mandatory to cite the author of this study as a co-author.

REFERENCES:
- [Background] El Fawal MH, Mohammed DA, Abou-Abbass H, Abbas M, Tamim H, Kanawati S. Laparoscopic Sleeve Gastrectomy under Awake Paravertebral Blockade Versus General Anesthesia: Comparison of Short-Term Outcomes. Obes Surg. 2021 May;31(5):1921-1928. doi: 10.1007/s11695-020-05197-6. Epub 2021 Jan 8. PMID 33417101
- [Background] Kanawati S, Fawal H, Maaliki H, Naja ZM. Laparoscopic sleeve gastrectomy in five awake obese patients using paravertebral and superficial cervical plexus blockade. Anaesthesia. 2015 Aug;70(8):993-5. doi: 10.1111/anae.13037. Epub 2015 Mar 10. PMID 25756905
- [Background] Subramani Y, Nagappa M, Wong J, Patra J, Chung F. Death or near-death in patients with obstructive sleep apnoea: a compendium of case reports of critical complications. Br J Anaesth. 2017 Nov 1;119(5):885-899. doi: 10.1093/bja/aex341. PMID 29077813
- [Background] Frey WC, Pilcher J. Obstructive sleep-related breathing disorders in patients evaluated for bariatric surgery. Obes Surg. 2003 Oct;13(5):676-83. doi: 10.1381/096089203322509228. PMID 14627460
- [Background] Beloeil H. Opioid-free anesthesia. Best Pract Res Clin Anaesthesiol. 2019 Sep;33(3):353-360. doi: 10.1016/j.bpa.2019.09.002. Epub 2019 Sep 26. PMID 31785720
- [Background] Gabriel RA, Swisher MW, Sztain JF, Furnish TJ, Ilfeld BM, Said ET. State of the art opioid-sparing strategies for post-operative pain in adult surgical patients. Expert Opin Pharmacother. 2019 Jun;20(8):949-961. doi: 10.1080/14656566.2019.1583743. Epub 2019 Feb 27. PMID 30810425
- [Background] Oderda GM, Senagore AJ, Morland K, Iqbal SU, Kugel M, Liu S, Habib AS. Opioid-related respiratory and gastrointestinal adverse events in patients with acute postoperative pain: prevalence, predictors, and burden. J Pain Palliat Care Pharmacother. 2019 Sep-Dec;33(3-4):82-97. doi: 10.1080/15360288.2019.1668902. Epub 2019 Oct 14. PMID 31609155
- [Background] Tashani OA, Astita R, Sharp D, Johnson MI. Body mass index and distribution of body fat can influence sensory detection and pain sensitivity. Eur J Pain. 2017 Aug;21(7):1186-1196. doi: 10.1002/ejp.1019. Epub 2017 Mar 6. PMID 28263427
- [Background] Phillips BT, Shikora SA. The history of metabolic and bariatric surgery: Development of standards for patient safety and efficacy. Metabolism. 2018 Feb;79:97-107. doi: 10.1016/j.metabol.2017.12.010. Epub 2018 Jan 5. PMID 29307519